CLINICAL TRIAL: NCT03369600
Title: Characterisation of Tissue Stiffness to Improve the Diagnosis and Management of Uterine Fibroids
Brief Title: Characterisation of Uterine Fibroid Tissue Stiffness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dr. Linda McLean (Other)
Collaborators: Ottawa Hospital Research Institute (Other); The Ottawa Hospital (Other)
Responsible Party: Sponsor-Investigator, Dr. Linda McLean, Co-Investigator, University of Ottawa
Organization: University of Ottawa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Protocol # 20170872-01H
Record Dates: First submitted 2017-11-29; First posted 2017-12-12 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Leiomyoma
Keywords: elastography
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Controls (Experimental): Women Supersonic Imagine Aixplorer SWE Ultrasound Imaging on two separate occasions.
  Interventions: Device: Supersonic Imagine Aixplorer SWE Ultrasound Imaging
- FIB-Sx (Experimental): Women receiving Supersonic Imagine Aixplorer SWE Ultrasound Imaging prior to elective hysterectomy for treatment of symptomatic uterine fibroids.
  Interventions: Device: Supersonic Imagine Aixplorer SWE Ultrasound Imaging
- FIB-Mx (Experimental): Women receiving Supersonic Imagine Aixplorer SWE Ultrasound Imaging prior to and at two points during elective medical therapy for treatment of symptomatic uterine fibroids.
  Interventions: Device: Supersonic Imagine Aixplorer SWE Ultrasound Imaging

INTERVENTIONS:
Device: Supersonic Imagine Aixplorer SWE Ultrasound Imaging — Consented women will attend 2+ sessions where they will be imaged using the Supersonic Imagine Aixplorer for Shear Wave Elastography imaging.

SUMMARY:
Uterine fibroids (leiomyomas, myomas, fibroids) are benign tumors of the uterus that can cause heavy menstrual bleeding, pain, and/or infertility. Fibroids can be managed with medication, surgery, or interventional radiology. While conservative methods that avoid surgical risks and complications are becoming more common, there are limitations to medical therapies including side effects, short durations of use, and incomplete response to treatment. To optimize patient outcomes, it is imperative clinicians and researchers better understand which patients may benefit from medical therapies and which may not. Fibroids with less blood supply can degenerate and take on a variety of histological characteristics (e.g. cystic, red, fatty, calcific) which may decrease response to medical management. These histological characteristics in degenerated fibroids correspond to altered mechanical properties, ranging from very soft to very hard. There is currently no guidance on how to predict medical responsiveness based on such fibroid characteristics. As a result, physicians treat patients empirically with medications, without the ability to counsel on effectiveness or failure rates. Our research goal is to understand if and how uterine fibroid tissue stiffness can predict response to medical therapies. To achieve this, the investigators will use a new ultrasound technology, called shear wave elastography (SWE), that non-invasively measures tissue stiffness and is currently used in practice for staging of chronic liver diseases; however, given that this technology is very new, evidence of its clinical application in gynecology is limited. Through implementing an innovative and multidisciplinary approach, the investigators will (1) systematically establish SWE as a feasible and reliable tool for measuring non-neoplastic myometrial and uterine fibroid tissue stiffness, and (2) use SWE to classify and monitor fibroid tissue properties in pre-menopausal women undergoing medical intervention for symptomatic uterine fibroids. Understanding the connection between pathological tissue properties and the success of medical therapies is essential to streamline assessment and intervention planning and improve overall patient outcomes for the many Canadian women who suffer from uterine fibroids.

DETAILED DESCRIPTION:
Aims and Objectives The goal of this project is to understand if and how uterine fibroid tissue stiffness, measured by SWE, can be used to predict and monitor response to medical therapy in patients with symptomatic uterine fibroids.

Aim 1: To assess the feasibility of using SWE for measuring stiffness of non-neoplastic myometrium and uterine fibroid tissue in pre-menopausal women Objective 1.1: Assess the inter- and intra-session reliability of measuring uterine tissue stiffness with SWE in 60 women with uterine fibroids and 60 healthy matched control participants.

Objective 1.2: Using data acquired from the 60 women with uterine fibroids, the validity of SWE will be assessed by comparing in vivo uterine tissue stiffness measured by SWE to the stiffness of surgically excised uterine tissue samples measured ex vivo by a mechanical tester.

Objective 1.3: To assess the confounding effect of age, parity, contraceptive use, and presence of fibroids on myometrial stiffness measured by SWE in 60 women with uterine fibroids and 60 healthy matched control participants.

Aim 2: To assess the clinical applicability of using tissue stiffness measured by SWE for the classification and monitoring of uterine fibroids in pre-menopausal women.

Objective 2.1: Determine if SWE is sensitive enough to identify differences in tissue stiffness between non-degenerative and degenerative fibroids, as validated by histology from surgically excised tissue samples of 60 women.

Objective 2.2: Determine if SWE is sensitive enough to identify differences in fibroid tissue stiffness in 60 women with uterine fibroids before and after two 3-month courses of SPRM therapy and evaluate if medical responsiveness (i.e. symptom relief) is related to baseline SWE measures.

Study Design: This will be a prospective case-control study that will used a mixed model (within and between subject) study design (Figure 1). Women with uterine fibroids and healthy matched control participants will be recruited and attend two or three US imaging sessions (depending on group assignment). Participants with fibroids will have both their myometrium and fibroid stiffness measured using SWE. Healthy matched controls will have their myometrium measured only. Participants with fibroids receiving surgical intervention will undergo a hysterectomy or myomectomy and tissue samples will be harvested and tested in a jig that measures stiffness under mechanical tension. Participants with fibroids seeking medical management will have an US imaging session before and after two 3-month courses of ulipristal acetate (UPA; an SPRM prescribed in Canada20).

Participants: Three groups of 60 premenopausal women over the age of 18 will be recruited:

1. Patients seeking surgical management for uterine fibroids (FIB-Sx) will be recruited from a list of patients consented for surgery (hysterectomy or myomectomy with primary indication of fibroids) by a member of The Ottawa Hospital Minimally Invasive Gynecology Group (led by Nominated Principal Applicant, S. Singh). FIB-Sx will be excluded if they have >5 fibroids identified on US or suspicion of leiomyosarcoma based on clinical, surgical, or gross pathological examination.
2. Patients seeking medical management for uterine fibroids (FIB-Mx) will be screened from a list of referrals to the Shirley E. Greenberg Women's Health Center (SEGWHC) at The Ottawa Hospital and recruited at the time of consult if they have been prescribed a course of UPA by their attending physician. FIB-Mx will be excluded if they have >5 fibroids identified on US or previous course of SPRM/GnRH analogues within 3 months of recruitment.
3. Healthy control participants (CON) (matched to FIB in age, parity, and BMI) will be recruited from the Ottawa community through advertisement posters, word of mouth, and social media. CON will be excluded is they have a history of uterine pathology (e.g. adenomyosis, hyperplasia, endometriosis), have irregular menstrual cycles, are currently pregnant or have been pregnant within the last six months prior to recruitment.

Initial assessment: Consented women in the control (CON) and surgical (FIB-Sx) streams will attend two evaluations. Consented women in the medical stream (FIB-Mx) will attend one visit at their earliest convenience after recruitment, another at three months after treatment initiation, and third visit at 6 months after treatment initiaition. At each visit, women will undergo shear wave elastography (SWE) and 3D US (Supersonic UltrafastTM Aixplorer®, Apexium Medical, Canada) assessments of their uterus as a whole, at 10 healthy sites and at up to 5 fibroid sites. SWE and volumes will be recorded in series of 10 frame clips. Morphologic measurements of the uterus and selected fibroids will be made and fibroids will be given identification numbers based on a 3D size and location map. SWE will be used to take relevant measures of tissue stiffness at all sites of interest. Three repetitions of each measurement will be performed. Women in the CON and FIB-Sx streams will receive a second identical imaging session during their first visit and a single imaging session during the second visit. Participants in the FIB-Mx stream will receive a single imaging session at each visit.

Surgical Intervention: the surgical approach (abdominal vs laparoscopic) will be recorded as well as secondary outcomes including operating time, blood loss, surgical technique conversions, failed/incomplete excisions, and additional procedures performed. These data will be used for descriptive purposes and contribute to the development of a database for our long-term research goal.

Tissue Sampling: For participants in the FIB-Sx stream, the surgical approach (myomectomy or hysterectomy + abdominal or laparoscopic), course of resection and secondary outcomes including operating time, blood loss, surgical technique, failed/incomplete excisions, intra- or post-operative complication and additional procedures will be recorded for descriptive purposes. Morcellated tissue specimens will be excluded. All surgically excised tissue will be sent to pathology for gross inspection and processing following standard procedures. For hysterectomy cases, a pathology assistant (trained and under the supervision of collaborator S. Strickland) will excise five 1cm3 samples of non-neoplastic tissue from myometrial sites-of interest and 1cm3 sections from each fibroid of interest. For myomectomy cases, 1cm3 sections from each fibroid of interest will similarly be excised. In surgical cases with >3 fibroids excised, the participating surgeon will include the study specific fibroid identification number given at the US imaging session in the pathology requisition. A member of the research team will meet the pathology assistant at the time of dissection to ensure each sample is placed in individual bottles with isotonic saline and labelled with its unique study identification number. Samples will be transported to M. Labrosse's (collaborator) laboratory at the Ottawa Heart Institute for mechanical testing.

Medical Intervention: Medical treatment will be recorded as well as secondary outcomes relating to patient symptoms and quality of life.These data will be used for descriptive purposes and contribute to the development of a database for our long-term research goal.

Mechanical Testing: All samples will be stored in saline and tested within 24 hours of excision. Samples will be further dissected into 2x10mm slices and loaded into a mechanical jig (Biotester, CellScale, Waterloo, Canada) at collaborator M. Labrosse's laboratory and tested at 37°C, cyclically in tension (1Hz, 2-3% strain) following procedures developed in the literature for mechanical testing on uterine tissue. The modulus of elasticity (E, kPa), analogous to stiffness, and stiffness contrast ratio (E_fibroid/E_myometrium ) will be calculated three times for each sample and averaged. The mechanical testing protocol will take approximately 2 hours to complete. Mechanical loading will be under displacement control (2-3% strain) to eliminate the risk damaging tissues, allowing for repeated measurements and histological analysis. All samples will be placed in 10% neutral buffered formalin immediately after testing and returned to pathology for definitive diagnosis. Pathology reports and slides will be retrospectively reviewed to extract descriptive fibroid characteristics. Members of the research team acquiring subsequent SWE measurements, mechanical stiffness measurements, and reviewing pathology reports will be blinded to results of initial SWE measurement.

Statistical analyses:All data will be tested for normality and equivalent non-parametric tests to those described below will be used as appropriate. All tests will be performed using SPSS statistical software (v25, IMB Corp., Armonk, USA) and significance will be accepted as p<0.05. Appropriate post-hoc comparisons will be performed. Dependent variables of SWE peak and mean stiffness are assumed to be interrelated.

Objective 1.1: Two-way (3x2) multivariate analyses of variance (MANOVAs) will test for significant differences in mean and peak stiffness (kPa) as they relate to the independent variable of test time (repetition and session) for each measurement site. One-way analyses of variance (ANOVAs) and dependent t-tests will be used for post-hoc Bonferroni corrected evaluation of significant main effects. Dependent t-tests will determine if measurement plane significantly affects SWE stiffness measures. Intra-class correlation coefficients and standard error of measurements will evaluate intra- and inter-session, and between-plane reliability of SWE stiffness measurements.

Objective 1.2: Univariate linear regressions will map the relationship between SWE mean and peak stiffness and the complex modulus of elasticity, with the complex modulus of elasticity considered the criterion standard. For non-linear relationships, appropriate transformations will be made.

Objective 1.3: Two-way multivariate analyses of covariance will test the effect of site (cervical junction, isthmus, fundus) and group (FIB vs CON) on peak and mean myometrial stiffness and the confounding effects of age, parity and contraceptive use on the adjusted group mean difference. Independent t-tests will be used for post-hoc evaluation if a significant main effect/interaction is observed. Logistic regressions will map the relationship of age, parity, and contraceptive use to myometrial stiffness at each measurement site. Acceptable regressions will explain >80% of the variance in the data. For non-linear relationships, appropriate transformations will be made.

Objective 2.1: Based on the pathology report, fibroids will be classified as either non-degenerative (i.e. normal) or degenerative (inclusive of all variations in presentation). One-way MANOVAs will evaluate between group differences in fibroid type (non-degenerative vs degenerative) and uterine tissue peak and mean stiffness measured with SWE, while post-hoc evaluation of significant main effects will involve independent t-tests using appropriate Bonferroni corrections.

Objective 2.2: SWE measurements will be ensemble averaged across intra-session repetitions for each site. Two-way MANOVAs will evaluate site and time (pre, post-course 1, post-course 2) differences in mean and peak stiffness measured with SWE One-way ANOVAs and dependant t-tests will be used for post-hoc Bonferroni corrected evaluation of significant main effects.

ELIGIBILITY:
Inclusion Criteria (All Participants)

* Age 18 or older
* Premenopausal
* No co-morbidities known to impact tissue properties

Inclusion (FIB-Sx and FIB-Mx groups)

* Diagnosis of fibroids by imaging (FIB-Mx and FIB-Sx groups)
* Scheduled to undergo hysterectomy (FIB-Sx) or medical therapy (FIB-Mx) to treat symptomatic uterine fibroids
* <6 fibroids identified by medical imaging

Inclusion (CON group)

* no known history of gynecological pathologies
* regular menstrual cycles

Exclusion Criteria (All Participants)

* confirmed or suspected uterine cancer
* pregnancy
* <6months post-partum
* history of caesarean delivery
* previous uterine surgery

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-17 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
In vivo Tissue Stiffness | 2 years
  Tissue stiffness measured by shear wave elastography and reported in kilopascals and m/s

SECONDARY OUTCOMES:
Ex vivo Tissue Stiffness | 2 years
  Tissue stiffness measured by mechanical uniaxial testing and reported in kilopascals
SWE Validity | 2 years
  Measures of tissue stiffness taken using shear wave imaging correlated to mechanical ex-vivo testing of tissues and assessed using correlations and/or linear regression.
SWE Reliability | 2 years
  Between- and within-session reliability of measures of tissue stiffness taken using shear wave imaging assessed using ICCs

CONTACTS AND LOCATIONS:
Overall Officials: Linda McLean, PhD, Principal Investigator — University of Ottawa; Sukhbir S Singh, MD, FRCSC, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- University of Ottawa, Motor Function Measurement Laboratory, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03369600/Prot_SAP_002.pdf